CLINICAL TRIAL: NCT01854723
Title: Basal Insulin Therapy in Patients With Insulin Resistance: A 6 Month Comparison of Insulin Glargine and NPH Insulin
Brief Title: Comparison Study of Insulin Glargine and NPH Insulin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-029B
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: Diabetes; Insulin glargine; NPH insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Isophane Insulin, Human; Insulin, Isophane; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Switching to NPH insulin (Experimental): Patients in this arm will be transitioned from insulin glargine to NPH insulin with subsequent titration according to algorithm within protocol. If needed, meal-time insulin will be added during study period.
  Interventions: Drug: Switching to NPH insulin
- Continuation of insulin glargine (Active Comparator): Patients in this arm will continue on insulin glargine and serve as a control group.
  Interventions: Drug: Continuation of insulin glargine

INTERVENTIONS:
Drug: Switching to NPH insulin — Patients in this arm will be transitioned from insulin glargine to NPH insulin with subsequent titration according to algorithm within protocol. If needed, meal-time insulin will be added during study period.
  Other Names: Humulin N; Novolin N; Novolin NPH; NPH Iletin II; Isophane insulin
  Arms: Switching to NPH insulin
Drug: Continuation of insulin glargine — Patients in this group will serve as a control group, and information will be collected regarding the safety, effectiveness, and cost of treatment for use in this study.
  Other Names: Lantus
  Arms: Continuation of insulin glargine

SUMMARY:
This study will compare the safety, effectiveness, and cost of two different types of long-acting insulin.

DETAILED DESCRIPTION:
In this study the investigators will be comparing two long-acting insulins, insulin glargine and NPH insulin. The trial will be evaluating differences in effectiveness, safety and cost between the two agents when used in patients on more than 80 units or 1unit/kg long-acting insulin. The investigators hypothesis is that patients switched from lantus to NPH will have improved blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at 22 Providence Medical Group primary care clinics
* Diagnosis of type 2 diabetes mellitus
* Currently using greater than 80 units/day of insulin glargine or greater than 1 unit/kg/day of insulin glargine
* Current A1C > 8.5% (within 3 months of randomization)

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Age > 85 years
* Self-reported history of severe hypoglycemia or hypoglycemia unawareness
* Hospice/limited life expectancy
* Current enrollment in Providence Medical Group Medication Assistance Program
* Current use of a GLP1 agonist (i.e., liraglutide, exenatide, exenatide extended-release)
* End stage renal disease (i.e., dialysis or estimated glomerular filtration rate <15 ml/min/1.73m2)
* Cirrhosis
* Unstable coronary artery disease or chronic heart failure (i.e. an exacerbation or hospitalization within 6 months pre-randomization)
* Psychiatric condition that prevents adequate follow-up (i.e., > 3 missed follow-up visits within a 3 month period or persistent non-adherence to dosing or monitoring recommendations)
* Active alcohol or drug abuse
* Inability to provide informed consent

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in A1C between groups at 6 months | 6 months

SECONDARY OUTCOMES:
Difference in A1C between groups at 3 months | 3 months
Difference in self-monitored blood glucose averages between groups | 6 months
  Outside of A1C, the investigators will also be comparing self-monitored blood glucose averages within each group and comparing them to one another.
Difference in incidence of hypoglycemia between each group | 6 months
  * Mild = symptoms consistent with hypoglycemia during which the subject was able to self-treat and was associated with blood glucose < 70mg/dL
  * Severe = symptoms consistent with hypoglycemia during which the subject required the assistance of another person and was associated with either a glucose level < 56 mg/dL or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon
  * Nocturnal hypoglycemia = hypoglycemia as described above occurring after the subject goes to bed and before the measurement of glucose, eating breakfast, or administration of any glucose-lowering agent in the morning
Difference in units of basal insulin used per day between groups | 6 months
Difference in total units of insulin per day between groups | 6 months
Difference in percent of patients who require initiation/titration of prandial insulin between each group | 6 months
Difference in rate of mortality in each group during study period | 6 months
Difference in morbidity between each group during study period | 6 months
  Morbidity defined as glycemia-related hospitalizations, ER visits, immediate care clinic visits (hypoglycemia, hyperglycemia, diabetic ketoacidosis, hyperosmolar hyperglycemic nonketotic syndrome, hospitalizations diagnosed as related to diabetes with diagnosis code)
Compare cost of insulin therapy over study period at study completion | 6 months
  Costs will be calculated as direct patient cost and total cost of medication.
Differences in change in weight during study period between groups | 6 months
  Weight change in each patient will be calculated using weight at study initiation and completion
Difference in number of visits with clinical pharmacist | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stephens, MD, Principal Investigator — Providence Medical Group
Locations (1):
- Providence Medical Group Northeast Clinic, Portland, Oregon, United States

REFERENCES:
- [Background] Wang Z, Hedrington MS, Gogitidze Joy N, Briscoe VJ, Richardson MA, Younk L, Nicholson W, Tate DB, Davis SN. Dose-response effects of insulin glargine in type 2 diabetes. Diabetes Care. 2010 Jul;33(7):1555-60. doi: 10.2337/dc09-2011. Epub 2010 Mar 31. PMID 20357371
- [Background] Fritsche A, Schweitzer MA, Haring HU; 4001 Study Group. Glimepiride combined with morning insulin glargine, bedtime neutral protamine hagedorn insulin, or bedtime insulin glargine in patients with type 2 diabetes. A randomized, controlled trial. Ann Intern Med. 2003 Jun 17;138(12):952-9. doi: 10.7326/0003-4819-138-12-200306170-00006. PMID 12809451
- [Background] Eliaschewitz FG, Calvo C, Valbuena H, Ruiz M, Aschner P, Villena J, Ramirez LA, Jimenez J; HOE 901/4013 LA Study Group. Therapy in type 2 diabetes: insulin glargine vs. NPH insulin both in combination with glimepiride. Arch Med Res. 2006 May;37(4):495-501. doi: 10.1016/j.arcmed.2005.10.015. PMID 16715577
- [Background] Yki-Jarvinen H, Kauppinen-Makelin R, Tiikkainen M, Vahatalo M, Virtamo H, Nikkila K, Tulokas T, Hulme S, Hardy K, McNulty S, Hanninen J, Levanen H, Lahdenpera S, Lehtonen R, Ryysy L. Insulin glargine or NPH combined with metformin in type 2 diabetes: the LANMET study. Diabetologia. 2006 Mar;49(3):442-51. doi: 10.1007/s00125-005-0132-0. Epub 2006 Feb 3. PMID 16456680
- [Background] Riddle MC, Rosenstock J, Gerich J; Insulin Glargine 4002 Study Investigators. The treat-to-target trial: randomized addition of glargine or human NPH insulin to oral therapy of type 2 diabetic patients. Diabetes Care. 2003 Nov;26(11):3080-6. doi: 10.2337/diacare.26.11.3080. PMID 14578243
- [Background] Massi Benedetti M, Humburg E, Dressler A, Ziemen M. A one-year, randomised, multicentre trial comparing insulin glargine with NPH insulin in combination with oral agents in patients with type 2 diabetes. Horm Metab Res. 2003 Mar;35(3):189-96. doi: 10.1055/s-2003-39080. PMID 12734781
- [Background] Rosenstock J, Schwartz SL, Clark CM Jr, Park GD, Donley DW, Edwards MB. Basal insulin therapy in type 2 diabetes: 28-week comparison of insulin glargine (HOE 901) and NPH insulin. Diabetes Care. 2001 Apr;24(4):631-6. doi: 10.2337/diacare.24.4.631. PMID 11315821
- [Background] Bota VM, Hirsch IB. Insulin glargine or neutral protamine Hagedorn in patients with severe insulin resistance: Is there a benefit? Endocr Pract. 2012 May-Jun;18(3):e49-51. doi: 10.4158/EP11302.CR. PMID 22232027